CLINICAL TRIAL: NCT06578416
Title: Developmental Trajectories to Stuttering Persistence and Recovery
Brief Title: The Development of Stuttering in Young Children
Status: Recruiting | Type: Observational
Sponsor: Michigan State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Bridget Walsh, Associate Professor of Communicative Sciences and Disorders, Michigan State University
Other Study IDs: 00001704; R01DC018000 (NIH)
Record Dates: First submitted 2024-08-01; First posted 2024-08-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Stuttering; Stuttering, Childhood; Stuttering, Developmental
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children who stutter: Preschool children who stutter aged 3 to 6-years
  Interventions: Diagnostic Test: Standardized assessments of speech and language abilities
- Children who do not stutter: Preschool children who do not stutter aged 4 to 6-years
  Interventions: Diagnostic Test: Standardized assessments of speech and language abilities

INTERVENTIONS:
Diagnostic Test: Standardized assessments of speech and language abilities — Standardized and observational assessment of speech and language abilities

SUMMARY:
The goal of this longitudinal research is to learn why some children "grow out" of stuttering, while others persist. Children who do and do not stutter aged 3-6 years are eligible to participate in our study. During the study, children's speech and language abilities will be assessed with standardized assessments, and they complete several child-friendly experiments. During these experiments, brain activity will be recorded using specialized caps while children describe pictures, children will speak in two virtual-reality scenarios, and produce speech while keeping to a beat.

DETAILED DESCRIPTION:
The length of participation in our study depends on the subset of activities completed. Families in the longitudinal study will take part in three visits each lasting approximately 2 hrs for up to 5 years.

Parents and caregivers will complete parent questionnaires (1 x each year for up to 5 years) and a 5-minute, online survey in between visits to the lab (1x each year for up to 5 years). Children will take part in standardized and observational assessments (1x each year for up to 5 years). These may cover aspects of social/emotional development, cognition, and speech, language, and hearing abilities. These tests are used to assess whether a child falls within or outside of the normative range for his/her age.

Children will participate in one or more of the following tasks (1x each year for up to 5 years)

* Listen to sounds or words and view or name pictures presented on a monitor. Brain activity electroencephalography (EEG) will be recorded while children listen to speech sounds and name pictures. This will be done with an elastic cap that holds special sensors (electrodes). Sensors will also be placed behind each ear, beside each eye, and under the left eye.
* Virtual reality (VR). Children wear a VR headset and experience virtual, age-appropriate talking situations (e.g., answering questions in a classroom). While they talk in these scenarios, the headset measures where they are looking (eye tracking), and sensors on their forehead, hand, and finger measure their heart rate and sweat response.
* Children will watch cartoons of animals jumping to a consistent beat (rhythm) and produce a word in time with the animal jumping/beat.
* Children will repeat nonwords, name pictures, or count while wearing a cap with sensors. Half of the sensors emit light through while the other half measures the reflected light. These sensors give us information about brain activity and are not harmful.

ELIGIBILITY:
Inclusion Criteria for controls:

* English as first/primary language
* No history of neurological disease
* Normal or corrected visual acuity
* No medications expected to affect performance
* No intellectual impairment, autism spectrum disorder, ADHD
* Age-appropriate scores on speech and language assessment battery
* Pass hearing screening at 20 dB at 500, 1000, 2000, and 4000, bilaterally

Inclusion Criteria for children who stutter:

* English as first/primary language
* No history of neurological disease
* Normal or corrected visual acuity
* No medications expected to affect performance
* No intellectual impairment or ASD Scores on speech and language assessments indicating stuttering, phonological (speech sound), or language disorders
* Pass hearing screening at 20 dB at 500, 1000, 2000, and 4000, bilaterally

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preschool children who do and do not stutter
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Stuttering Severity | 1 x each year for up to 5 years
  Assess speech for the presence of stuttering disfluencies and calculate the severity of stuttering based on parent ratings and calculated as the percentage of disfluent syllables out of the total syllables of speech produced.
Virtual reality speaking scenarios | 1 x each year for up to 5 years
  Record looking events in msec during virtual reality scenarios (classroom of children and kitten)
Virtual reality speaking scenarios | 1 x each year for up to 5 years
  Pulse oximetry measures will be taken with a photoplethysmograph transducer (Biopac TSD200) secured around the distal phalanx of the fourth finger of the child's non-dominant hand with a Velcro strap. Two measures will be analyzed. (1) Blood pulse volume (BPV) amplitude, the average trough-to-peak amplitude (in volts) of pulse cycles across segments where the child is producing speech and (2) Pulse rate (PR in pulses per minute ppm), will be recorded for each speech segment then averaged. These pulse oximetry measures will be taken during the viewing of virtual reality scenarios (classroom of children and kitten)
Virtual reality speaking scenarios | 1 x each year for up to 5 years
  Electrodermal (skin conductance) recordings will be collected from the hands while children are immersed in virtual reality speaking scenarios (classroom of children and kitten). We report skin conductance levels and skin conductance response frequency and amplitude in microSiemens (mS).
EEG recording of event-related brain potentials | 1 x each year for up to 5 years
  Electroencephalographic (EEG) recordings of event-related brain potentials will be conducted during a picture identification task. ERPs will be averaged across conditions and reported in microvolts.
Speech production synchronization | 1 x each year for up to 5 years
  We record productions of a word spoken to the beat under different feedback conditions. We will assess timing measures reflecting the accuracy with which children synchronize their speech to the beat and retain the rhythm.
fNIRS recording of cortical hemodynamic responses | 1 x each year for up to 5 years
  Cerebral hemodynamic responses are recorded during the experiment with a continuous-wave fNIRS system (NIRx, Inc). The system uses LED light source optodes, and avalanche photodiode optode detectors for measuring intensity changes in the diffused light at a 10-Hz sampling rate. The optodes are embedded in a standard EEG cap. The concentrations of oxygenated hemoglobin and deoxygenated hemoglobin in micromols will be calculated across trial intervals as participants describe child-friendly picture scenes. These responses will then be averaged across trials for each child.

CONTACTS AND LOCATIONS:
Locations (1):
- Developmental Speech Lab, East Lansing, Michigan, United States